CLINICAL TRIAL: NCT06892327
Title: BIOmetric MEasurements in Diagnostics: Comparison of EXperts and IA-assisted Residents
Acronym: BIOMEDEXIA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2025_001
Record Dates: First submitted 2025-03-12; First posted 2025-03-24 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy
Keywords: ultrasound; Biometric measurements; artificial intelligence; obstetrics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Routine Follow-Up: Patients scheduled for a standard biometric ultrasound.: Maternal Age: Pregnant women aged between 18 and 45 years. Pregnancy Type: Singleton viable pregnancy (excluding twin or multiple gestations).
  Gestational Age: Between 17 weeks and 38 weeks of gestation.
  Interventions: Other: standard biometric ultrasound

INTERVENTIONS:
Other: standard biometric ultrasound — In this study, biometric measurements were systematically performed for each patient using both manual methods and an artificial intelligence (AI) system (Live View Assist, Samsung). The AI system provided real-time guidance by identifying anatomical landmarks and assisting in the measurement of key biometric parameters, including Femur Length (FL), Abdominal Circumference (AC), Head Circumference (HC), and Biparietal Diameter (BPD). This dual approach ensured that both manual and AI-assisted methods were applied uniformly as part of routine clinical care.

SUMMARY:
Obstetric ultrasound is the cornerstone of fetal growth assessment. It provides essential biometric measurements for estimating fetal weight, monitoring growth and identifying conditions such as intrauterine growth retardation (IUGR) or macrosomia. The accuracy of these measurements depends largely on the expertise of the operator. Experienced practitioners excel at positioning the probe, identifying anatomical landmarks and obtaining reproducible measurements. In contrast, novice operators, such as medical residents, may find it difficult to capture optimal images or identify precise landmarks, resulting in significant variability. This inter-observer variability, well documented even among experts, can have an impact on clinical decisions and obstetric management. For novices, variability is more pronounced, which can affect diagnostic reliability and patient care. Improving resident training is therefore essential to reduce this variability. Traditional solutions to minimizing variability, such as increased supervision, face limitations due to time constraints and resource availability. Recent advances in Artificial Intelligence (AI) could help in the training of residents. In obstetrics, AI could potentially automate biometric measurements by identifying key anatomical landmarks and performing precise, consistent measurements. These systems might standardize acquisition and reduce variability, making measurements less dependent on operator experience. AI technologies could significantly improve novice performance by potentially shortening the learning curve and enhancing measurement reliability. This might enable residents to work more independently while maintaining accuracy. Despite these potential advantages, few studies would have rigorously compared AI-assisted novice performance with that of expert practitioners under real-world conditions.This study aims to assess the possible effectiveness of AI in supporting novice operators during obstetric biometric measurements. The primary objective would be to determine whether AI assistance could enable novices to achieve measurement accuracy comparable to that of experienced practitioners, while potentially improving reproducibility and reducing inter-observer variability.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged between 18 and 40 years.
* Singleton or twin ongoing pregnancies.
* Gestational age between 20 and 36 weeks of amenorrhea (WA).
* Patients scheduled for a biometric ultrasound (standard follow-up).

Exclusion Criteria:

* Known major fetal anomalies that could affect biometric measurements.
* Technical difficulties during the ultrasound (e.g., maternal obesity, complex abdominal scars).
* History of severe maternal conditions affecting biometric measurements (e.g., uterine malformations)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant woman
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of biometric measurements: Assessment of agreement between manual and AI-assisted measurements. | 36 weeks amenorrhea
  The individual biometric measurements, such as biparietal diameter (BPD), head circumference (HC), abdominal circumference (AC), and femur length (FL), will be presented separately based on their respective units (cm).
  The estimated fetal weight, which will be based on the aggregation of these various measurements (BPD, HC, AC, FL), will be reported in kilograms (kg). This estimate will be calculated using fetal growth formulas adapted to these parameters.
  We will clarify that the fetal weight estimate will be calculated based on a model that incorporates these different measurements in the appropriate units.
  In summary, each measurement will be clearly separated based on its unit, and the fetal weight estimate will be explained to show how the different measurements are combined.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Maternité Croix Rousse, Lyon, France